CLINICAL TRIAL: NCT05447052
Title: The Biomimetic Stent and Vascular Functions Study-The MIMICS FLOW STUDY
Brief Title: The Biomimetic Stent and Vascular Functions Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Chistos Rammos, Prof. Dr. med. C. Rammos, MD, FESC, MHBA, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The MIMICS FLOW STUDY
Record Dates: First submitted 2022-06-02; First posted 2022-07-07 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bio-MIMICS Stent (Experimental): Helical shaped BioMimics 3D Stent
  Interventions: Device: Bio-MIMICS 3D Stent
- Innova Stent (Active Comparator): Conventional: Nitinol Stent
  Interventions: Device: Innova Stent

INTERVENTIONS:
Device: Bio-MIMICS 3D Stent — Bio-MIMICS Stent implantation
  Arms: Bio-MIMICS Stent
Device: Innova Stent — Innova Stent implantation
  Arms: Innova Stent

SUMMARY:
The aim of this IIT is to determine the potential improvement and impact of the BioMimics 3D Stent System in the SFA on local vascular function.

DETAILED DESCRIPTION:
The MIMICS FLOW Study is a single-center, single-blind, investigator-initiated, randomized parallel group trial.

The impact of a novel biomimetical stent with a helical curvature provides superior hemodynamic and biomechanical performance and advantages. Additionally, it promotes swirling blood flow, elevating wall sheer strength, which is patency-protective and might impact on vascular functions due to completely different vascular properties through altered blood flow.

The influence of the novel devices and stent-platforms with improved hemodynamic capabilities with respect to vasomotor of the vessel wall, vascular function and vascular compliance can be measured by FMD, arterial stiffness indices and vascular strain analysis.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral artery disease
* Target lesions in the proximal (3 cm distal to the CFA-bifurcation) middle and distal SFA
* Clinical diagnosis of chronic, symptomatic lower limb ischemia as defined by Rutherford 2,3,4
* Planed peripheral intervention TASC A-D
* Subject must be between 18 and 85 years old
* Female of childbearing potential must have a negative pregnancy test within 10 days prior to index procedure and utilize reliable birth control until completion of the 12 month angiographic evaluation
* Vessel diameter >/= 4.0 mm and </=7.0 mm
* Target lesion length < 140 mm (segment to be stented)
* Willing to comply with the specified follow-up evaluation
* Written informed consent prior to any study procedures
* Pretreatment with an adequately sized ballon (1:1 ration to nonstenotic vessel diameter)
* usage of Biomimics stent as described in the IFU, especially regarding stent diameters and vessel size

Exclusion Criteria:

* Bifurcational lesions of the CFA and lesions including the first 3 cm of the SFA, due to technical aspects of FMD measurement
* Requiring stent implantation in the PA
* Instent-Restenosis
* Thrombolysis within 72 Hours prior to the index procedure
* Aneurysm formations in the femoral artery or popliteal artery
* Concomitant hepatic insufficiency, deep venous thrombus, coagulation disorder or receiving immunosuppressant therapy
* Unstable angina pectoris at the time of the enrollment
* Recent myocardial infarction or stroke <30 days prior to the index procedure
* Life expectancy less than 12 months
* Septicaemia at the time of enrollment
* Known or suspected active infection at the time of the index procedure, excluding an infection of a lower extremity wound of the target limb
* Known or suspected allergies or contraindications to aspirin, clopidogrel or heparin
* Presence of other hemodynamically significant outflow lesions in the target limb requiring a planned surgical intervention or endovascular procedure within 30 days after the index procedure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-04-26 (Estimated); Study Completion 2025-04-26 (Estimated)

PRIMARY OUTCOMES:
Change of flow-mediated vasodilation (FMD) of the nonstenotic segment of the proximal SFA after procedure | 1 month
  FMD represents the percent diameter gain as calculated based on preischemia and postischemia diameter measurements of the femoral artery.
Change of flow-mediated vasodilation (FMD) of the nonstenotic segment of the proximal SFA after procedure | 12 months
  FMD represents the percent diameter gain as calculated based on preischemia and postischemia diameter measurements of the femoral artery.

SECONDARY OUTCOMES:
Changes in pulse wave velocity | Baseline, followed at 1 and 12 months
  Changes in cardiovascular function measured by pulse wave velocity in m/s
Changes in augmentation index | Baseline, followed at 1 and 12 months
  Changes in cardiovascular function measured by augmentation index in %
Changes in vascular strain | Baseline, followed at 1 and 12 months
  Changes in cardiovascular function measured by vascular strain in %
Changes in peripheral perfusion determined by ABI (ankle brachial index) | Baseline, followed at 1 and 12 months
  ABI measurements are conducted using a Doppler probe on tibial and anterior artery locations. The highest value will be used for calculation and divided by the highest systolic brachial Doppler pressure
Primary patency (PP) of target lesion | Baseline, followed at 1 and 12 months
  Primary patency determined by PVR measurement with ultrasound
Changes in clinical symptoms | Baseline, followed at 1 and 12 months
  Clinical symptoms of patients determined by Walking impairment questionaire (WIQ)
Changes in six-minute walk test | Baseline, followed at 1 and 12 months
  Six-minute walk test determined by pain-free walking distance in m
Freedom from Target Lesion Revascularization | Baseline, followed at 1 and 12 months
  Freedom from Target Lesion Revascularization (FTLR)
Number of participants with treatment-related adverse events | Baseline, followed at 1 and 12 months
  Number of participants with treatment-related adverse events as assessed by SDWS
Changes of inflammatory profile measured by hs-CRP in mg/dl | Baseline, followed at 1 and 12 months
  Blood samples are collected at the below mentioned time points
Changes of inflammatory profile measured by oxLDL in µg/l | Baseline, followed at 1 and 12 months
  Blood samples are collected at the below mentioned time points
Changes of inflammatory profile measured by Interleukin-6 in pg/ml | Baseline, followed at 1 and 12 months
  Blood samples are collected at the below mentioned time points

CONTACTS AND LOCATIONS:
Overall Officials: Christos Rammos, Professor, Principal Investigator — University Hospital, Essen
Locations (1):
- University of Essen, Clinic of Cardiology and Angiology, Essen, North Rhine-Westphalia, Germany